CLINICAL TRIAL: NCT03571789
Title: Carotid Artery Implant for Trapping Upstream Emboli for Preventing Stroke in Atrial Fibrillation Patients
Acronym: CAPTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javelin Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CL-150
Record Dates: First submitted 2018-05-30; First posted 2018-06-28 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation
Keywords: AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, non-randomized, open-label, first-in-human (FIH) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vine™ implantation bilaterally in the common carotid arteries (Experimental): Vine™ is a permanent carotid filter made from a single nitinol wire. It is configured to capture emboli exceeding 1.2mm in size, which originate in the heart and large arteries below the neck. Vine™ has a helical structure, with leading and supporting coils interposed by a filter section.
  Interventions: Device: Vine™

INTERVENTIONS:
Device: Vine™ — The Vine™ is made of a super-elastic nitinol wire comprises a helix that resides within the CCA lumen and a linear stem that traverses the CCA wall. The helix includes three segments: supporting coils, filter, and leading coils.
  The device is available in sizes of 6.0mm - 10.0mm (in 0.5mm intervals) to accommodate individual CCA diameters

SUMMARY:
Vine™ is a permanent carotid filter designed to provide protection against embolic stroke in people with atrial fibrillation. It is implanted bilaterally in the common carotid arteries from a thin needle under ultrasound guidance. The procedure is performed without general anesthesia and takes minutes. The safety, feasibility and tolerability of Vine™ will be evaluated. Patients who are eligible will receive Vine™ and will be followed-up for a year after device implantation.

DETAILED DESCRIPTION:
CAPTURE is a prospective, single-arm, multicenter trial, designed to evaluate the safety, feasibility and tolerability of the Vine™ permanent carotid filter. The trial will enroll up to 30 patients, and will be conducted in up to five sites worldwide. All enrolled patients will be invited for non-invasive follow-up tests and clinical evaluations according to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Atrial fibrillation (AF): documented persistent or permanent
2. CHA2DS2-VASc score ≥ 4
3. Age > 50
4. Unsuitable for oral anticoagulation therapy (OAC), defined as contraindicated for OAC, patient refusing OAC, or physician is reluctant to prescribe OAC
5. Maximal (systolic) CCA diameter range: ≥ 5.3mm and ≤ 9.8mm
6. CCA accessibility: up to 60mm from skin to CCA center, safe approach
7. Patient is willing to provide informed consent
8. Patient is willing to complete all scheduled follow-up

Exclusion Criteria:

1. Evidence of carotid stenosis > 30% [CCA, internal carotid artery (ICA), or external carotid artery (ECA)
2. Evidence of any atherosclerotic disease in CCA above the clavicles
3. Evidence of carotid dissection
4. Pre-existing stent(s) in CCA
5. Contraindicated or allergic to antiplatelet therapy, or any medication required during the study
6. Recent stroke, TIA, or myocardial infarction (MI) within two months prior to index procedure
7. Female who is pregnant or who is planning to become pregnant during the course of the study
8. Life expectancy of less than 1 year
9. Active systemic infection
10. Known sensitivity to nickel or titanium metals, or their alloys
11. Known hereditary or acquired coagulation disorders
12. Any planned surgical or endovascular procedure within 14 days prior to or 30 days after the index procedure
13. A co-morbid disease or condition that could confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments
14. Current use or a recent history of illicit drug(s) use or alcohol abuse (defined as regular or daily consumption of more than four alcoholic drinks per day)
15. Active participation in another investigational drug or device treatment study
16. Any other condition that in the opinion of the investigator may adversely affect the safety of the subject or would limit the subject's ability to complete the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with no incidence of device and/or procedure related Major Adverse Events (MAEs) | 30 days from implantation procedure
  Major Adverse Events (MAEs) are defined as:
  * Death
  * Major and minor strokes
  * Major bleeding
  * Common carotid artery (CCA) stenosis > 70%
  * Vine™ migration
  * CCA thrombus
  * Any complications in the CCA requiring endovascular treatment or surgery
Number of patients with Procedure Success | 30 days from implantation procedure
  Procedure Success is defined as Proper Vine™ Position in each CCA
  Proper Vine™ Position is defined as:
  * Supporting coil in contact with artery walls
  * No migration
  * No fracture
  * No Vine™ coils or portions thereof visible outside the arterial lumen
  * No entangled or overlapping coils

SECONDARY OUTCOMES:
Number of patients with no incidence of device and/or procedure related Major Adverse Events (MAEs) | within 3, 6, months,1, 2, 3, 4 and 5 years of implantation procedure
  Death
  * Major and minor strokes
  * Major bleeding
  * Common carotid artery (CCA) stenosis > 70%
  * Vine™ migration
  * CCA thrombus
  * Any complications in the CCA requiring endovascular treatment or surgery
Number of Successful Delivery and Deployment Attempts | within 4 hours of implantation procedure
  Successful Delivery and Deployment Attempts is defined as Proper Vine™ Position
Number of patients with properly positioned Vine™ in each CCA | within 3, 6, months,1, 2, 3, 4 and 5 years of implantation procedure
  Proper implant position

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, Principal Investigator — Na Homolca Hospital; Jan Van der Heijden, MD, Principal Investigator — St. Antonius Hospital; Tom De Potter, MD, Principal Investigator — OLV Ziekenhuis; Stefan Verheye, MD, Principal Investigator — ZNA Stuivenberg
Locations (4):
- Belgium (2):
  - OLV Ziekenhuis, Aalst
  - ZNA Stuivenberg, Antwerp
- Na Homolce Hospital, Prague, Czechia
- Sint-Antonius ziekenhuis, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy VY, Neuzil P, de Potter T, van der Heyden J, Tromp SC, Rensing B, Jiresova E, Dujka L, Lekesova V. Permanent Percutaneous Carotid Artery Filter to Prevent Stroke in Atrial Fibrillation Patients: The CAPTURE Trial. J Am Coll Cardiol. 2019 Aug 20;74(7):829-839. doi: 10.1016/j.jacc.2019.04.035. Epub 2019 May 11. PMID 31085320